CLINICAL TRIAL: NCT07164794
Title: A Prospective Study of Memantine Hydrochloride for the Treatment of Prostate Cancer Patients
Brief Title: Memantine Hydrochloride in Prostate Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bin Xu (Other)
Collaborators: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor-Investigator, Bin Xu, Researcher, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZDSYLL297-P01
Record Dates: First submitted 2025-08-13; First posted 2025-09-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC); Prostate Cancer; Neuroendocrine Prostate Cancer (NEPC)
Keywords: Memantine; mCRPC; Prospective Study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Memantine Hydrochloride (Experimental): Participants will receive the study drug, memantine hydrochloride, in addition to their ongoing standard of care treatment. The standard of care background therapy consists of Androgen Deprivation Therapy (ADT) using a GnRH agonist or antagonist , combined with a novel endocrine therapy such as abiraterone acetate or enzalutamide, based on the patient's prior treatment history.
  The dosing for memantine hydrochloride is as follows:
  Week 1: 5 mg once daily. Week 2: 10 mg once daily. Week 3: 15 mg once daily. Week 4 and thereafter: 20 mg once daily as a maintenance dose.
  Interventions: Drug: Memantine Hydrochloride

INTERVENTIONS:
Drug: Memantine Hydrochloride — Memantine Hydrochloride is administered orally, once daily, in combination with the patient's ongoing standard of care treatment for metastatic castration-resistant prostate cancer (mCRPC).
  The dosing follows a weekly titration schedule for the first three weeks to reach the maintenance dose.
  Week 1: 5 mg once daily. Week 2: 10 mg once daily. Week 3: 15 mg once daily. Week 4 and onwards: 20 mg once daily. This intervention is being studied to evaluate its potential to reduce neuroendocrine differentiation and correct castration resistance in advanced prostate cancer.

SUMMARY:
The goal of this clinical trial is to learn if long-term use of memantine hydrochloride can treat, prevent, or correct castration resistance and drug resistance in advanced prostate cancer. The study will enroll male patients aged 18 and older diagnosed with metastatic castration-resistant prostate cancer (mCRPC) who have previously failed first or second-line treatments. The main questions it aims to answer are:

What is the progression-free survival (PFS) in patients treated with memantine hydrochloride? What is the disease control rate (DCR) and what is the change in Prostate-Specific Antigen (PSA) levels after treatment?

Researchers will compare outcomes from participants in this single-arm study to an external historical control group of patients who received traditional treatment to see if the addition of memantine hydrochloride improves prognosis.

Participants will be asked to do the following:

Continue their standard of care treatment, which includes Androgen Deprivation Therapy (ADT) and a novel endocrine therapy.

Take the study drug, memantine hydrochloride, with the dose gradually increasing over the first three weeks to a maintenance dose.

Attend regular follow-up appointments for blood tests to check PSA levels and undergo imaging scans to monitor the disease status. These follow-ups will occur one month after starting the drug and every three months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with metastatic castration-resistant prostate cancer (mCRPC) who have failed one or two prior lines of therapy. Patients with concomitant Alzheimer's disease will be prioritized for enrollment.
3. Complete clinical baseline data must be available, and the patient must be willing to undergo long-term follow-up.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

Exclusion Criteria:

1. Patients with metastatic prostate cancer at initial diagnosis who have not progressed to mCRPC.
2. Patients with a concurrent primary malignancy at another site.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Assessed at 1 month post-treatment initiation, and every 3 months thereafter, until disease progression, death, or study completion, up to a maximum of 1 year
  PFS is defined as the time from treatment initiation to the first documentation of disease progression or death from any cause, whichever comes first. Disease progression is a composite event, defined by either biochemical progression (per PCWG3 criteria using blood PSA levels) or radiological progression (per RECIST 1.1 criteria using imaging such as pelvic CT or prostate MRI).

IPD SHARING:
Plan to Share IPD: Yes
After the publication of primary study results in a peer-reviewed journal, de-identified individual participant data (IPD) that underlie the results, as well as the study protocol, will be made available upon reasonable request to the Principal Investigator (PI).

DOCUMENTS (2):
  • Study Protocol (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT07164794/Prot_000.pdf
  • Informed Consent Form (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT07164794/ICF_001.pdf